CLINICAL TRIAL: NCT02528227
Title: NICU Parent Education Program
Acronym: NICU PEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Elisabeth McGowan, Assistant Professor of Pediatrics, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 12-0074
Record Dates: First submitted 2015-08-05; First posted 2015-08-19 (Estimated); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Language Development; Premature Infant; Neurodevelopmental Outcomes
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Language Curriculum (Experimental): The Language Intervention group will receive some of the known methods for early language development. Six lessons will include: Knowing your Baby, Reading Aloud, Sing-A-Long, Mimicking First Sounds, Language Game and Narrating Your Day. Parents will receive feedback every 2 weeks from a Language Environment Analysis digital language processor (LENA).
  Interventions: Other: Know Your Baby Language Curriculum; Other: Reading Aloud Language Curriculum; Other: Sing A Long Language Curriculum; Other: Mimicking First Sounds Language Curriculum; Other: Language Games and Narrating Your Day Language Curriculum
- Health and Safety Curriculum (Placebo Comparator): Parents will receive six lessons on important infant safety topics including, feeding safety, care seat safety, bath safety, back to sleep/SIDS prevention, taking a temperature and signs of infection, infection control methods and vaccine information. Parents will receive LENA feedback at discharge from NICU.
  Interventions: Other: Feeding Safety; Other: Car Seat Safety; Other: Bath Safety; Other: Back to Sleep/SIDS prevention; Other: Taking a Temperature and Signs of Infection; Other: Infection Control Measures and Vaccine Information

INTERVENTIONS:
Other: Know Your Baby Language Curriculum — Early language activities that parents can do with their infants
  Arms: Language Curriculum
Other: Reading Aloud Language Curriculum — Early language activity that parents can do with their infants
  Arms: Language Curriculum
Other: Sing A Long Language Curriculum — Early language activity that parents can do with their infants
  Arms: Language Curriculum
Other: Mimicking First Sounds Language Curriculum — Early language activity that parents can do with their infants
  Arms: Language Curriculum
Other: Language Games and Narrating Your Day Language Curriculum — Early language activity that parents can do with their infants
  Arms: Language Curriculum
Other: Feeding Safety — Part of Health and Safety Curriculum
  Arms: Health and Safety Curriculum
Other: Car Seat Safety — Part of Health and Safety Curriculum
  Arms: Health and Safety Curriculum
Other: Bath Safety — Part of Health and Safety Curriculum
  Arms: Health and Safety Curriculum
Other: Back to Sleep/SIDS prevention — Part of Health and Safety Curriculum
  Arms: Health and Safety Curriculum
Other: Taking a Temperature and Signs of Infection — Part of Health and Safety Curriculum
  Arms: Health and Safety Curriculum
Other: Infection Control Measures and Vaccine Information — Part of Health and Safety Curriculum
  Arms: Health and Safety Curriculum

SUMMARY:
The purpose of this study is to adminster one of two education programs to parents of preterm infants in the NICU to evaluate language and cognitive outcomes of their infants.

DETAILED DESCRIPTION:
The long term goal of this research is to determine the language environment necessary in the NICU for very preterm infants to optimize their long-term language and cognitive development. This study will pilot an early language intervention with parents of preterm infants in the NICU the purpose of which is to provide a structured curriculum for the family to guide their language interactions with their infant. The aim is to increase the adult word counts and conversational turns in the NICU and to improve Bayley III language and cognitive scores at 12 months and 24 months corrected age.

The hypotheses is that increasing early language exposure in the NICU will result in improved lanugage and cognitive scores. The investigators plan on testing the hypothesis by the following specific aims.

1. Determine the effectiveness of a structured language curriculum with parents of preterm infants in the NICU on increasing the amount of early language exposure.
2. Test the the hypothesis that increased early language exposure will result in higher Bayley III language and cognitive scores.

ELIGIBILITY:
Inclusion Criteria:

* Receiving care at Women & Infants' Hospital NICU,
* Providence RI gestational age 23 - 32 weeks,
* RI resident

Exclusion Criteria:

* Unable to understand or speak English,
* congenital or chromosomal disorder likely to affect cognitive or speech development,
* parental loss of custody

Ages: 23 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2013-01; Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Bayley III cognitive composite score | 24 months
  Bayley III cognitive score (mean 100, standard deviation 15)
Bayley III language composite score | 24 months
  Bayley III Language score (mean 100, standard deviation 15)
Bayley III Expressive Language Score | 24 months
  Bayley III Expressive Language (mean 10, standard deviation 3)
Bayley III Receptive Language Score | 24 months
  Bayley III Receptive Language (mean 10, standard deviation 3)
Bayley III Motor Composite score | 24 months
  Bayley III Motor composite score (mean 100, standard deviation 15)

SECONDARY OUTCOMES:
Infant vocalizations Count | 32 weeks post menstrual age
  LENA recordings of infant vocalizations (software derived recording of all speech related sounds recorded in a 16 hour time period).
Infant vocalizations Count | 34 weeks post menstrual age
  LENA recordings of infant vocalizations (software derived recording of all speech related sounds recorded in a 16 hour time period).
Infant vocalizations Count | 36 weeks post menstrual age
  LENA recordings of infant vocalizations (software derived recording of all speech related sounds recorded in a 16 hour time period).
Conversational turns Count | 32 weeks post menstrual age
  LENA recordings of infant-parent conversational turns (softward derived recording of adult-child interactions that estimates the number of reciprocal vocalizations between infant and adult within 5 seconds, and recorded for a 16 hour time period).
Conversational turns Count | 34 weeks post menstrual age
  LENA recordings of infant-parent conversational turns (softward derived recording of adult-child interactions that estimates the number of reciprocal vocalizations between infant and adult within 5 seconds, and recorded for a 16 hour time period).
Conversational turns Count | 36 weeks post menstrual age
  LENA recordings of infant-parent conversational turns (softward derived recording of adult-child interactions that estimates the number of reciprocal vocalizations between infant and adult within 5 seconds, and recorded for a 16 hour time period).
Adult word count Count | 32 weeks post menstrual age
  LENA recordings of adult word count (softward derived number of adult words spoken during a 16 hour period).
Adult word count | 34 weeks post menstrual age
  LENA recordings of adult word count (softward derived number of adult words spoken during a 16 hour period).
Adult word count | 36 weeks post menstrual age
  LENA recordings of adult word count (softward derived number of adult words spoken during a 16 hour period).
Bayley III cognitive composite score | 12 month
  Bayley III cognitive score (mean 100, standard deviation 15)
Bayley III motor composite score | 12 month
  Bayley III motor score (mean 100, standard deviation 15)
Bayley III expressive language score | 12 month (mean 10, standard deviation 3)
  Bayley III expressive language score (mean 100, standard deviation 15)
Bayley III receptive language score | 12 month (mean 10, standard deviation 3)
  Bayley III receptive language score (mean 100, standard deviation 15)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth C McGowan, MD, Principal Investigator — Women and Infants' Hospital Providence RI
Locations (1):
- Women and Infants' Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Result] Caskey M, Stephens B, Tucker R, Vohr B. Importance of parent talk on the development of preterm infant vocalizations. Pediatrics. 2011 Nov;128(5):910-6. doi: 10.1542/peds.2011-0609. Epub 2011 Oct 17. PMID 22007020
- [Result] Caskey M, Stephens B, Tucker R, Vohr B. Adult talk in the NICU with preterm infants and developmental outcomes. Pediatrics. 2014 Mar;133(3):e578-84. doi: 10.1542/peds.2013-0104. Epub 2014 Feb 10. PMID 24515512
- [Derived] McGowan EC, Caskey M, Tucker R, Vohr BR. A Randomized Controlled Trial of a Neonatal Intensive Care Unit Language Intervention for Parents of Preterm Infants and 2-Year Language Outcomes. J Pediatr. 2024 Jan;264:113740. doi: 10.1016/j.jpeds.2023.113740. Epub 2023 Sep 16. PMID 37717908